CLINICAL TRIAL: NCT02684357
Title: BI 655066 Versus Ustekinumab and Placebo Comparators in a Randomized Double Blind trIal for Maintenance Use in Moderate to Severe Plaque Type Psoriasis-2 (UltIMMa-2)
Brief Title: BI 655066 Versus Placebo & Active Comparator (Ustekinumab) in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M15-995; 2015-003622-13 (EudraCT Number); 1311.28 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-02-16; First posted 2016-02-18 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Part A) (Placebo Comparator): Participants were randomized to receive double-blind (DB) placebo by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: placebo for risankizumab; Drug: placebo for ustekinumab
- Ustekinumab (Part A) (Active Comparator): Participants randomized to receive double-blind (DB) ustekinumab 45 or 90 mg (based on screening weight) by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: ustekinumab; Drug: placebo for risankizumab
- Risankizumab (Part A) (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: risankizumab; Drug: placebo for ustekinumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab pre-filled syringe, administered by subcutaneous (SC) injection
  Other Names: BI 655066; ABBV-066; SKYRIZI
  Arms: Risankizumab (Part A)
Drug: ustekinumab — Ustekinumab pre-filled syringe, administered by subcutaneous (SC) injection
  Arms: Ustekinumab (Part A)
Drug: placebo for risankizumab — Placebo for risankizumab pre-filled syringe, administered by subcutaneous (SC) injection
  Arms: Placebo (Part A); Ustekinumab (Part A)
Drug: placebo for ustekinumab — Placebo for ustekinumab pre-filled syringe, administered by subcutaneous (SC) injection
  Arms: Placebo (Part A); Risankizumab (Part A)

SUMMARY:
This is a randomized double blind, double dummy, placebo and active comparator controlled, parallel design study that is being performed to assess the safety and efficacy of risankizumab (BI 655066) to support registration for the treatment of moderate to severe chronic plaque psoriasis in adult patients.

DETAILED DESCRIPTION:
Participants were randomized to receive either placebo, ustekinumab, or risankizumab in Part A. All participants received 2 sets of injections to maintain the blind: the placebo arm received placebo for risankizumab and placebo for ustekinumab), the risankizumab arm received risankizumab and placebo for ustekinumab, and the ustekinumab arm received ustekinumab and placebo for risankizumab. Participants who received placebo in Part A switched to risankizumab in Part B; participants who received ustekinumab or risankizumab in Part A continued to receive the same treatment (ustekinumab or risankizumab) in Part B.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per International Council on Harmonisation (ICH) M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

  *Women of childbearing potential are defined as:
  * having experienced menarche and are
  * not postmenopausal (12 months with no menses without an alternative medical cause) and are
  * not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).
* Age ≥ 18 years at screening
* Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug.Duration of diagnosis may be reported by the patient,
* Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomization):

  1. Have an involved body surface area (BSA) ≥ 10% and
  2. Have a Psoriasis Area and Severity Index (PASI) score ≥ 12 and
  3. Have a static Physician Global Assessment (sPGA) score of ≥ 3.
* Must be candidates for systemic therapy or phototherapy for psoriasis treatment, as assessed by the investigator
* Must be a candidate for treatment with Stelara® (ustekinumab) according to local label.
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practices (GCP) and local legislation

Exclusion criteria:

* Patients with:

  1. non-plaque forms of psoriasis (including guttate, erythrodermic, or pustular),
  2. current drug-induced psoriasis (including an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium),
  3. active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis that might confound trial evaluations according to investigator's judgment,
* Previous exposure to BI 655066,
* Currently enrolled in another investigational study or less than 30 days (from screening) since completing another investigational study (participation in observational studies is permitted),
* Previous exposure to ustekinumab (Stelara®),
* Use of any restricted medication, or any drug considered likely to interfere with the safe conduct of the study,
* Major surgery performed within 12 weeks prior to randomization or planned within 12 months after screening (e.g., hip replacement, aneurysm removal, stomach ligation),
* Known chronic or relevant acute infections including active tuberculosis, HIV or viral hepatitis; QuantiFERON® tuberculosis (TB) test or purified protein derivative (PPD) skin test will be performed according to local labelling for comparator products. If the result is positive, patients may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment should have been initiated and maintained according to local country guidelines,
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix,
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and electrocardiogram [ECG]), or laboratory value at the screening visit outside the reference range that is in the opinion of the investigator, is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data,
* History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients,
* Women who is pregnant, nursing, or who plans to become pregnant while in the trial,
* Previous enrolment in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Background] Sonenshein GE, Siekevitz M, Siebert GR, Gefter ML. Control of immunoglobulin secretion in the murine plasmacytoma line MOPC 315. J Exp Med. 1978 Jul 1;148(1):301-12. doi: 10.1084/jem.148.1.301. PMID 97359
- [Derived] Strober B, Armstrong A, Rubant S, Patel M, Wu T, Photowala H, Crowley J. Switching to risankizumab from ustekinumab or adalimumab in plaque psoriasis patients improves PASI and DLQI outcomes for sub-optimal responders. J Dermatolog Treat. 2022 Nov;33(7):2991-2996. doi: 10.1080/09546634.2022.2095328. Epub 2022 Jul 31. PMID 35839335
- [Derived] Lebwohl MG, Soliman AM, Yang H, Wang J, Hagan K, Padilla B, Pinter A. Impact of Risankizumab on PASI90 and DLQI0/1 Duration in Moderate-to-Severe Psoriasis: A Post Hoc Analysis of Four Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Feb;12(2):407-418. doi: 10.1007/s13555-021-00660-3. Epub 2021 Dec 18. PMID 34921669
- [Derived] Augustin M, Lambert J, Zema C, Thompson EHZ, Yang M, Wu EQ, Garcia-Horton V, Geng Z, Valdes JM, Joshi A, Gordon KB. Effect of Risankizumab on Patient-Reported Outcomes in Moderate to Severe Psoriasis: The UltIMMa-1 and UltIMMa-2 Randomized Clinical Trials. JAMA Dermatol. 2020 Dec 1;156(12):1344-1353. doi: 10.1001/jamadermatol.2020.3617. PMID 33052382
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118
- [Derived] Gordon KB, Strober B, Lebwohl M, Augustin M, Blauvelt A, Poulin Y, Papp KA, Sofen H, Puig L, Foley P, Ohtsuki M, Flack M, Geng Z, Gu Y, Valdes JM, Thompson EHZ, Bachelez H. Efficacy and safety of risankizumab in moderate-to-severe plaque psoriasis (UltIMMa-1 and UltIMMa-2): results from two double-blind, randomised, placebo-controlled and ustekinumab-controlled phase 3 trials. Lancet. 2018 Aug 25;392(10148):650-661. doi: 10.1016/S0140-6736(18)31713-6. Epub 2018 Aug 7. PMID 30097359
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 577 subjects were enrolled; 86 subjects failed screening and are excluded from the analyses.
Groups:
- Placebo (Part A): Participants randomized to receive double-blind (DB) placebo by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
- Placebo/Risankizumab (Part B): Participants randomized to receive placebo in Part A switched to risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Ustekinumab/Ustekinumab (Part B): Participants randomized to receive ustekinumab in Part A continued to receive ustekinumab 45 mg or 90 mg (based on screening weight) by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Risankizumab/Risankizumab (Part B): Participants randomized to receive risankizumab in Part A continued to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
Period: Part A
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Started | 98 | 99 | 294 | 0 | 0 | 0
Completed | 94 | 96 | 292 | 0 | 0 | 0
Not Completed | 4 | 3 | 2 | 0 | 0 | 0
Not completed — Adverse Event (Worsening of Disease) | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Started | 0 | 0 | 0 | 94 (Participants who received placebo in Part A received risankizumab in Part B) | 94 (2 participants who received ustekinumab in Part A did not receive a dose of study drug in Part B.) | 291 (1 participant who received risankizumab in Part A did not receive a dose of study drug in Part B)
Completed | 0 | 0 | 0 | 91 | 90 | 278
Not Completed | 0 | 0 | 0 | 3 | 4 | 13
Not completed — Adverse Event (Other) | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Total
Number analyzed (Participants) | 98 | 99 | 294 | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.26) | 48.6 (14.81) | 46.2 (13.68) | 46.7 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 91 | 155
  Male | 67 | 66 | 203 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 12 | 44 | 75
  Not Hispanic or Latino | 79 | 87 | 250 | 416
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 7 | 4 | 25 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 2 | 2 | 10 | 14
  White | 87 | 91 | 255 | 433
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Non-responder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 2.0 | 74.8
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata (baseline weight [≤100 kg vs >100 kg] and prior exposure to tumor necrosis factor [TNF] antagonists [0 vs ≥1]). If there was a stratum containing zero count, 0.1 was added to each cell; Adjusted percentage difference = 72.5, 95% CI 2-sided [66.8 to 78.2] — 95% CI for adjusted difference of 2 treatment groups, calculated from the Cochran-Mantel-Haenszel test adjusted for the comparison of 2 treatment groups. If there was a stratum containing zero count, 0.1 was added to each cell

2. Primary Outcome: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 5.1 | 83.7
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 78.5, 95% CI 2-sided [72.4 to 84.5] — 95% CI for adjusted difference of 2 treatment groups, calculated by the Cochran-Mantel-Haenszel test adjusted for the comparison of 2 treatment groups. If there was a stratum containing zero count, 0.1 was added to each cell

3. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 3.1 | 51.0
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 47.5, 95% CI 2-sided [40.9 to 54.2] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 2.0 | 50.7
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 48.2, 95% CI 2-sided [41.9 to 54.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 0 to 30, where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired. A 5-point change from baseline is considered a clinically important difference. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 4.1 | 66.7
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 62.2, 95% CI 2-sided [55.5 to 68.9] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Symptom Scale (PSS) Score of 0 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 0 | 31.3
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 31.2, 95% CI 2-sided [25.7 to 36.6] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Achieving PASI90 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 47.5 | 74.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 27.6, 95% CI 2-sided [16.7 to 38.5] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 61.6 | 83.7
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 22.3, 95% CI 2-sided [12.0 to 32.5] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI00 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 24.2 | 50.7
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 27.0, 95% CI 2-sided [17.0 to 37.0] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 25.3 | 51.0
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 26.3, 95% CI 2-sided [16.1 to 36.4] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants Achieving PASI90 at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 7
Time Frame: Week 52
Population: ITT population. Non-responder imputation. Analysis performed on all participants randomized to ustekinumab or risankizumab treatment in Part A.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 99 | 294
percentage of participants | 50.5 | 80.6
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 30.2, 95% CI 2-sided [19.6 to 40.9] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 9
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 99 | 294
percentage of participants | 30.3 | 59.5
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 29.5, 95% CI 2-sided [18.9 to 40.1] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 99 | 294
percentage of participants | 30.3 | 59.5
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 29.5, 95% CI 2-sided [18.9 to 40.1] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 12 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 69.7 | 88.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 19.2, 95% CI 2-sided [9.5 to 28.8] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 12 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 64.6 | 82.3
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 18.0, 95% CI 2-sided [7.8 to 28.3] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 5
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 99 | 294
percentage of participants | 46.5 | 66.7
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 20.2, 95% CI 2-sided [9.1 to 31.4] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Change From Baseline to Week 16 in PSS Total Score in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. A negative change in PSS total score indicates improvement. Last observation carried forward (LOCF) imputation was used for missing data.
Time Frame: Week 16
Population: ITT population. Last observation carried forward. Participants randomized to placebo or risankizumab with an observed baseline PSS and at least one post-baseline PSS observation on or prior to Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 85 | 227
units on a scale | -0.027 (0.3316) | -6.402 (0.2193)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); P-value calculated by the van Elteren test stratified for baseline weight (≤100 kg vs >100 kg) and prior exposure to TNF antagonists (0 vs ≥1); Test type: Other; p < 0.001, van Elteren test; Mean Difference (Final Values) = -6.375, 95% CI 2-sided [-7.102 to -5.648]

18. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: as for outcome 14
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 98 | 294
percentage of participants | 6.1 | 90.8
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 84.7, 95% CI 2-sided [79.0 to 90.4] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 99 | 294
percentage of participants | 54.5 | 83.3
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 29.1, 95% CI 2-sided [18.5 to 39.6] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 14
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 99 | 294
percentage of participants | 76.8 | 91.5
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 14.7, 95% CI 2-sided [5.9 to 23.5] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of study drug (up to 55 weeks).
Description: TEAEs and TESAEs in Part A are defined as events from the first dose of study drug in Part A until prior to the first dose in Part B (Week 16) or up to 105 days after the last dose of study drug if the participant discontinued in Part A; AEs in Part B are defined as events from the first dose of study drug in Part B (Week 16) until up to 105 days after the last dose of study drug.
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/99 | 1/294 | 0/94 | 0/94 | 1/291
Serious Adverse Events (participants affected / at risk) | 1/98 | 3/99 | 6/294 | 4/94 | 3/94 | 13/291
Other Adverse Events (participants affected / at risk) | 8/98 | 14/99 | 29/294 | 27/94 | 26/94 | 67/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=98) | Ustekinumab (Part A) (N=99) | Risankizumab (Part A) (N=294) | Placebo/Risankizumab (Part B) (N=94) | Ustekinumab/Ustekinumab (Part B) (N=94) | Risankizumab/Risankizumab (Part B) (N=291)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=98) | Ustekinumab (Part A) (N=99) | Risankizumab (Part A) (N=294) | Placebo/Risankizumab (Part B) (N=94) | Ustekinumab/Ustekinumab (Part B) (N=94) | Risankizumab/Risankizumab (Part B) (N=291)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (6) | 3 (3) | 2 (2) | 3 (3) | 6 (6)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 6 (6) | 2 (2) | 5 (7) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 11 (11) | 9 (13) | 8 (8) | 24 (28)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 10 (10) | 17 (22) | 14 (16) | 34 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.